CLINICAL TRIAL: NCT06001957
Title: Genetic Background Assessment With Whole Exome Sequencing in a Giant Coronary Artery Ectasia: a Pilot Study.
Brief Title: Whole Exome Sequencing in Coronary Artery Ectasia
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Collaborators: Medical University of Warsaw (Other); Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Konrad Stępień, Principal Investigator, MD, Assistant, Jagiellonian University
Other Study IDs: 1072.6120.49.2022
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Coronary Ectasia; Coronary Aneurysm
Keywords: Coronary ectasia; Coronary aneurysm; Whole exome sequencing; Mutations
MeSH Terms: conditions — Coronary Aneurysm | interventions — Exome; Genetic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from proband was obtained from peripheral blood and extracted using standard protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Proband: Patient with extremely giant coronary artery ectasia (CAE) and positive family history
  Interventions: Diagnostic Test: Whole exome sequencing

INTERVENTIONS:
Diagnostic Test: Whole exome sequencing — Bioinformatic analysis of raw WES data and variants prioritization were performed as previously described.
  Reads were aligned to the hg38 reference genome sequence and visualized by Integrative Genomic Viewer.
  Other Names: Genetic analysis

SUMMARY:
The goal of this observational study is to assess the role of the whole exome sequencing (WES) application in patients with giant coronary artery ectasia (CAE) with a high-risk of genetic background.

The main question it aims to answer are:

* the assessment of role of WES in CAE
* the detection of novel pathogenic mutations associated with CAE development

DETAILED DESCRIPTION:
Coronary artery aneurysm and ectasia (CAAE) is defined as a dilation of the coronary artery by at least 1.5 times compared to the adjacent segment. The incidence of CAAE is reported in 0.3-5.3% of patients undergoing coronary angiography. Giant CAAE is a rare phenomenon characterized by a dilation of a coronary artery exceeding 2 to 4 centimeters and it was found only in 0.02% of patients undergoing coronary angiography.

The most common etiology of CAAE is atherosclerosis, followed by Kawasaki disease, infectious septic emboli, connective tissue disease and arteritis. Iatrogenic causes are less common.

There are few genetic reports on potential loci associated with CAAE. Meta-analysis of genome wide association studies performed in European and Japanese population of children with Kawasaki disease has identified ITPKC, FCGR2A, CASP3 and FAM167A genomic regions to be associated with susceptibility to develop CAAE. Furthermore, 9p21 variant has been linked with coexistence of coronary artery disease, cerebral artery aneurysms and aortic aneurysms, mainly due to suspected potential adverse vascular remodeling. Nevertheless, the direct association of specific genetic variants with CAAE formation, especially with those giants, has not been proven.

Therefore, the investigators aim to assess the role of the whole exome sequencing (WES) application in patients with giant coronary artery ectasia (CAE) with a high-risk of genetic background.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed giant coronary artery aneurysm and ectasia (CAAE)
* high risk of genetic background

Exclusion Criteria:

* the lack of informed consent for whole exome sequencing (WES) analysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with extremely giant coronary artery ectasia (CAE) and positive family history.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
The novel pathogenic mutations associated with CAE development | Until June 11, 2023
  Reads of WES will be aligned to the hg38 reference genome sequence and visualized by Integrative Genomic Viewer.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Coronary Disease and Heart Failure, John Paul II Hospital in Krakow, Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No